CLINICAL TRIAL: NCT01681602
Title: Preserving Quality of Life, Physical Health and Functional Ability in Alzheimer's Disease: The Effect of Physical Exercise
Brief Title: Effect of Physical Exercise in Alzheimer Patients
Acronym: ADEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steen G Hasselbalch, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-3-2011-128
Record Dates: First submitted 2012-04-30; First posted 2012-09-10 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Exercise; Cognition; Quality of life; Cardiovascular fitness; Behavioural or psychological symptoms; Physical fitness
MeSH Terms: conditions — Alzheimer Disease; Motor Activity | interventions — Exercise; Endurance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): 16 weeks of aerobic exercise
  Interventions: Other: Aerobic exercise
- Control group (No Intervention): Usual care.

INTERVENTIONS:
Other: Aerobic exercise — Physical exercise in the intervention group will be delivered as an individually tailored program consisting of 4 weeks of adaptation exercise followed by 12 weeks of continuously supervised moderate aerobic exercise 1 hour three times a week. The participants can choose from treadmill, stationary bike and crosstrainer.
  Other Names: Endurance training
  Arms: Intervention group

SUMMARY:
Background: Current treatment for Alzheimer's disease (AD) is symptomatic and can only temporarily slow down progression.

Exercise has the potential to improve cognition, psychological symptoms, physical performance and quality of life, but evidence is scarce. Previous trials are short, often underpowered and involving home based light exercise programs. Most have included nursing homes residents with severe or undefined dementia. The aim of the ADEX trial is to establish whether exercise is effective in improving cognition, physical performance and quality of life as well as reducing the prevalence of psychological symptoms among AD patients.

Methods: The ADEX Trial is a multicentre, single-blind, randomized clinical trial. Based on power calculations the investigators plan to recruit 192 home-dwelling patients aged 50-90 years with mild to moderate AD. The participants will be randomly allocated into two groups: An intervention group attending 16 weeks of continuously supervised moderate aerobic exercise 1 hour three times a week and a control group only receiving usual care. The hypothesis is that aerobic exercise will improve physical function, the cognitive and daily functioning and quality of life in people with mild to moderate AS.

Blood sampling will be performed in all subjects to examine effects on biomarkers. A subgroup of the patients will also undergo MRI, PiB-PET and lumbar puncture to investigate structural changes and β-amyloid accumulation.

Further, a health-economic analysis will be performed.

Recruitment was started in January 2012. Last study visits are planned to be performed in January 2014 and results will be available in 2014. This RCT will contribute to evidence regarding the potential effects of a systematic program of physical exercise for patients with Alzheimer's disease.

DETAILED DESCRIPTION:
see protocol article

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are (table 1)
* Age between 50 and 90 years
* A score of 20 or more on the Mini Mental State Examination (MMSE)
* Imaging (CT or MR of cerebrum) consistent with AD
* Have a caregiver with regular contact to the participant (more than once a month) who is also willing to participate in the study
* In general good health allowing the participant to participate in physical exercise.
* At least 7 years of schooling and Danish speaking
* Visual acuity and hearing must permit neuropsychological testing.
* If the patient is receiving anti-dementia medication or mood stabilizing medication, these must have been given in stable doses for at least 3 months.

Exclusion Criteria:

* Participation in aerobic exercise (moderate to hard intensity) more than 2 times a week on a regular basis.
* Any musculoskeletal or joint impairment that could interfere with completion of the study (significant joint problems, back pain or pain in arms and legs that provide problems with mobility in daily activities)
* Male participants with a combination of two or more of the following risk factors even if asymptomatic: smokers, hypertension and hypercholesterolemia
* Major neurologic (other than AD), cardiac or other medical diseases that constitutes a contraindication to physical activity. Stent operation or previous myocardial infarction is not an exclusion criteria if the participant has had a recent (within 3 months) normal exercise tests .
* Severe cerebro vascular disease judged from the CT or MR scans and remarkable hypertension defined as Systolic blood pressure >180 and diastolic >100
* Severe psychiatric disease, as well as alcohol or drug abuse within the last 2 years

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Symbol Digit Modalities Test | Change in score from baseline to 16 weeks

SECONDARY OUTCOMES:
NPI (psychological symptoms.) | Change in score from baseline to 16 weeks
Astrand submaximal bicycle test for estimating VO2 max | Change in score from baseline to 16 weeks
Euro-qol-5D-5L (health related quality of life) | Change in score from baseline to 16 weeks
Alzheimer's disease Assessment Scale - Cognitive section (ADAS-cog). | Change in score from baseline to 16 weeks
Changes in physical fitness | Change in score from baseline to 16 weeks
  Timed up and go test (TUG), 10 m walk, 10m Dual-Task, 400m fast walking, Sit-to-stand (number in 30 sec.)(STS).
Self-efficacy scale | Change in score from baseline to 16 weeks
Verbal fluency | Change in score from baseline to 16 weeks
Stroop | Change in score from baseline to 16 weeks
MMSE (Mini Mental State Examination) | Change in score from baseline to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steen G Hasselbalch, Professor, Principal Investigator — Memory Disorders Research Group, Department of Neurology, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Danish Dementia Research Centre, Department of Neurology, Rigshospitalet., Copenhagen, Copenhagen Ø, Denmark

REFERENCES:
- [Derived] Delgado-Peraza F, Nogueras-Ortiz C, Simonsen AH, Knight DD, Yao PJ, Goetzl EJ, Jensen CS, Hogh P, Gottrup H, Vestergaard K, Hasselbalch SG, Kapogiannis D. Neuron-derived extracellular vesicles in blood reveal effects of exercise in Alzheimer's disease. Alzheimers Res Ther. 2023 Sep 20;15(1):156. doi: 10.1186/s13195-023-01303-9. PMID 37730689
- [Derived] Frederiksen KS, Jensen CS, Hogh P, Gergelyffy R, Waldemar G, Andersen BB, Gottrup H, Vestergaard K, Wermuth L, Sondergaard HB, Sellebjerg F, Hasselbalch SG, Simonsen AH. Aerobic exercise does not affect serum neurofilament light in patients with mild Alzheimer's disease. Front Neurosci. 2023 Jan 24;17:1108191. doi: 10.3389/fnins.2023.1108191. eCollection 2023. PMID 36761410
- [Derived] Musaeus CS, Johansen LB, Hasselbalch S, Beyer N, Hogh P, Siebner HR, Frederiksen KS. Sixteen Weeks of Aerobic Exercise does not Alter Resting-state Connectivity of the Precuneus in Patients with Alzheimer's Disease. Curr Alzheimer Res. 2022;19(2):171-177. doi: 10.2174/1567205019666220304091241. PMID 35249488
- [Derived] Clemmensen FK, Hoffmann K, Siersma V, Sobol N, Beyer N, Andersen BB, Vogel A, Lolk A, Gottrup H, Hogh P, Waldemar G, Hasselbalch SG, Frederiksen KS. The role of physical and cognitive function in performance of activities of daily living in patients with mild-to-moderate Alzheimer's disease - a cross-sectional study. BMC Geriatr. 2020 Nov 27;20(1):513. doi: 10.1186/s12877-020-01926-9. PMID 33246408
- [Derived] Frederiksen KS, Larsen CT, Hasselbalch SG, Christensen AN, Hogh P, Wermuth L, Andersen BB, Siebner HR, Garde E. A 16-Week Aerobic Exercise Intervention Does Not Affect Hippocampal Volume and Cortical Thickness in Mild to Moderate Alzheimer's Disease. Front Aging Neurosci. 2018 Sep 25;10:293. doi: 10.3389/fnagi.2018.00293. eCollection 2018. PMID 30319397
- [Derived] Sopina E, Sorensen J, Beyer N, Hasselbalch SG, Waldemar G. Cost-effectiveness of a randomised trial of physical activity in Alzheimer's disease: a secondary analysis exploring patient and proxy-reported health-related quality of life measures in Denmark. BMJ Open. 2017 Jun 14;7(6):e015217. doi: 10.1136/bmjopen-2016-015217. PMID 28615271